CLINICAL TRIAL: NCT04058782
Title: Impact of Peripheral Vascular Stiffness Assessment on Risk Prediction in Patients With Myocardial Infarction
Acronym: RIGID-MI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Fédération Française de Cardiologie (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018_43; 2018-A03276-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-08-07; First posted 2019-08-16 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Myocardial Infarction; Vascular Stiffness; Heart Failure
Keywords: Prognosis; Vascular stiffness; Heart failure; Myocardial infarction
MeSH Terms: conditions — Myocardial Infarction; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample for total blood, plasma and peripheral blood mononuclear cell collection at 1-month.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with myocardial
  Interventions: Other: Imaging evaluation for vascular assessment

INTERVENTIONS:
Other: Imaging evaluation for vascular assessment — At 1month after MI, Blood sample for total blood, plasma and PBMC collection, ECG, 3D-trans thoracic echocardiography for ventriculo-arterial coupling assessment, Vascular doppler for peripheral artery disease assessment, Arterial stiffness evaluation, Bilateral transcranial doppler for HITS evaluation

SUMMARY:
Risk assessment after myocardial infarction is critical in daily practice and evolution toward heart failure especially diastolic heart failure remains a key issue. All consecutive patients with myocardial infarction (either STEMI or NSTEMI but excluding type 2 MI) presenting at university hospital of Lille within 48 hours after symptom onset will be recruited in the RIGID-MI registry. The RIGID-MI study proposes to deeply evaluate at 1 month after MI: peripheral vascular disease, vascular stiffness, ventriculo-arterial coupling and other usual risk factors. The main objective is to identify clinical, biological and imaging parameters associated with poor prognosis, especially evolution toward diastolic heart failure, recurrence of MI, and bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Affiliated to national health insurance (French social security number)
* Presenting with MI within 48 hours of symptom onset

Exclusion Criteria:

* Patient under curatorship
* Type 2 MI
* Presenting with MI after 48 hours of symptom onset
* Pregnancy or lactating
* Refuse to participate
* No national health insurance (No French social security number)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with myocardial infarction (either STEMI or NSTEMI but excluding type 2 MI) presenting at university hospital of Lille within 48 hours after symptom onset will be recruited in the RIGID-MI registry.
  Over a 5-year period of time from 2019 to 2024. Planned population of 2000 patients. Follow-up every year by visit or phone contact up to 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-02-17 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
MACE: Major adverse cardiovascular events | at 5 years
  A composite of cardiovascular death, ischemic stroke, myocardial infarction, systemic embolism, acute limb ischemia, coronary revascularization, hospitalization for heart failure

SECONDARY OUTCOMES:
Cardiovascular death | at 5 years
Myocardial infarction | at 5 years
Ischemic stroke | at 5 years
Systemic embolism | at 5 years
Acute limb ischemia | at 5 years
Coronary revascularization | at 5 years
Hospitalization for heart failure | at 5 years
All-cause death | at 5 years
Bleeding as assessed by Bleeding Academic Research Consortium (BARC) | at 5 years
Bleeding as assessed by GUSTO Bleeding Criteria | at 5 years
  Global Utilization Of Streptokinase And Tpa For Occluded Arteries (GUSTO) definition for bleeding range to 1. Severe or Life-threatening/ 2. Moderate/ 3. Mild
Bleeding as assessed by Thrombolysis in Myocardial Infarction (TIMI) criteria | at 5 years
Bleeding as assessed by ISTH definitions | at 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Lemesle, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Institut Coeur-Poumon, CHU, Lille, France